CLINICAL TRIAL: NCT01596777
Title: Effects of 500 mg Immediate Release and Extended Release Methylnaltrexone on Loperamide-induced Delay of the Oro-cecal and Whole-gut Transit Time in Healthy Subjects
Acronym: LOP-MNTX-2009
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: LOP-MNTX-2009
Record Dates: First submitted 2012-05-07; First posted 2012-05-11 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Intestinal Obstruction
Keywords: Loperamide-induced obstipation; Methylnaltrexone; oro-cecal transit time; whole gut transit time; Pharmacokinetics
MeSH Terms: conditions — Intestinal Obstruction | interventions — Loperamide; methylnaltrexone; Sulfasalazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A (Placebo Comparator): Administration of LOP placebo (-24 h, -12 h, -1 h, 12 h), Colon Transit (-24 h, -12 h, -1 h), SSP (+ 2 h) and MNTX placebo (0 h). To asses the oro-cecal and whole-gut transit time under placebo condition.
  Interventions: Drug: Loperamide placebo; Drug: Methylnaltrexone placebo; Device: Colon Transit; Drug: Sulfasalazine
- Treatment B (Placebo Comparator): Administration of LOP 4 mg (-24 h, -12 h, -1 h, 12 h), Colon Transit (-24 h, -12 h, -1 h), SSP (+ 2 h) and MNTX placebo (0 h). To asses the oro-cecal and whole-gut transit time under loperamide-induced obstipation condition.
  Interventions: Drug: Loperamide; Drug: Methylnaltrexone placebo; Device: Colon Transit; Drug: Sulfasalazine
- Treatment C (Active Comparator): Administration of LOP 4 mg (-24 h, -12 h, -1 h, 12 h), Colon Transit (-24 h, -12 h, -1 h), SSP (+ 2 h) and MNTX 12 mg sc. (0 h). To assess the effects of methylnaltrexone in preventing loperamide-induced delay of the oro-cecal and whole-gut transit time and to measure pharmacokinetics of methylnaltrexone after subcutaneous administration.
  Interventions: Drug: Loperamide; Drug: Methylnaltrexone 12 mg sc.; Device: Colon Transit; Drug: Sulfasalazine
- Treatment D (Active Comparator): Administration of LOP 4 mg (-24 h, -12 h, -1 h, 12 h), Colon Transit (-24 h, -12 h, -1 h), SSP (+ 2 h) and MNTX IR (0 h). To assess the effects of methylnaltrexone in preventing loperamide-induced delay of the oro-cecal and whole-gut transit time and to measure pharmacokinetics of methylnaltrexone after oral administration of immediate release capsule.
  Interventions: Drug: Loperamide; Drug: Methylnaltrexone IR capsule; Device: Colon Transit; Drug: Sulfasalazine
- Treatment E (Active Comparator): Administration of LOP 4 mg (-24 h, -12 h, -1 h, 12 h), Colon Transit (-24 h, -12 h, -1 h), SSP (+ 2 h) and MNTX ER (0 h). To assess the effects of methylnaltrexone in preventing loperamide-induced delay of the oro-cecal and whole-gut transit time and to measure pharmacokinetics of methylnaltrexone after oral administration of extended release capsule.
  Interventions: Drug: Loperamide; Drug: Methylnaltrexone ER capsule; Device: Colon Transit; Drug: Sulfasalazine

INTERVENTIONS:
Drug: Loperamide — 20 ml Loperamid-ratiopharm® Lösung (ratiopharm) in 180 ml apple juice prepared before administration
  Other Names: LOP 4 mg
  Arms: Treatment B; Treatment C; Treatment D; Treatment E
Drug: Loperamide placebo — 200 ml apple juice
  Other Names: LOP placebo
  Arms: Treatment A
Drug: Methylnaltrexone placebo — Methylnaltrexone placebo capsule (identical to MNTX IR and MNTX ER)
  Other Names: MNTX placebo
  Arms: Treatment A; Treatment B
Drug: Methylnaltrexone 12 mg sc. — RELISTOR 12 mg/0.6 ml Injektionslösung (Wyeth)
  Other Names: MNTX 12 mg sc.
  Arms: Treatment C
Drug: Methylnaltrexone IR capsule — Methylnaltrexone bromide 500 mg IR capsule
  Other Names: MNTX IR
  Arms: Treatment D
Drug: Methylnaltrexone ER capsule — Methylnaltrexone bromide 500 mg ER capsule
  Other Names: MNTX ER
  Arms: Treatment E
Device: Colon Transit — 3x1 capsules containing radio-opaque marker of 6 different shapes (in two consecutive study periods, capsules with different shapes of the markers are given)
Drug: Sulfasalazine — 500 mg Azulfidine® (Pharmacia)
  Other Names: SSP

SUMMARY:
The purpose of this study is to describe the effects of methylnaltrexone in preventing loperamide-induced delay of the oro-cecal and whole-gut transit time and measure pharmacokinetics of methylnaltrexone after subcutaneous and oral administration of immediate release and extended release capsules.

DETAILED DESCRIPTION:
The increasing prevalence of opioid use and consequently, opioid-induced bowel dysfunction has prompted interest in identifying effective treatment options. Until now, the treatment of opioid-induced constipation (OIC) has been viewed as an extension of constipation in general. Traditional therapies for constipation such as bulking agents, stool softeners, stimulant laxatives, and osmotic agents are commonly utilized, but the effects of such therapies are nonspecific and are often generating diarrhea or cramps and some of these drugs cause severe side effects. Furthermore, these conventional measures are sometimes insufficient in some patients, especially those requiring increasing doses of opioids.

Opioid-induced constipation is predominantly mediated by gastrointestinal μ-opioid receptors. Selective blockade of these peripheral receptors might relieve constipation without compromising centrally mediated effects of opioid analgesia or precipitating withdrawal.

Naloxone is a competitive antagonist of opioid receptors inside and outside the central nervous system used as a solution for injection in the treatment of opioid overdose. When administered orally, it can reduce opioid-induced constipation due to a local action in the gut.

Another way to prevent central actions is the use of opioid antagonists which can't penetrate the blood-brain barrier such as methylnaltrexone and alvimopan. Their antagonism of μ-opioid receptors in the gastrointestinal tract seems to reverse opioid-induced gut hypomotility.

It is assumed that methylnaltrexone after oral administration influences intestinal motility by local blockade of opioid receptors along the luminal surface of the gut. Because methylnaltrexone seems to have an absorption window in the proximal small intestine as caused by lower activity of P-glycoprotein in that region (similar to other quaternary compounds, eg. trospium chloride), immediate release (uncoated) methylnaltrexone is better absorbed form the small intestine and might therefore be less active than the enteric-coated drug.

However, the pharmacokinetic and pharmacodynamic data on oral methylnaltrexone are very preliminarily so far. Furthermore, intestinal transit time has been measured using lactulose as a probe compound that has an own laxative effect.

Therefore, the following clinical study was initiated to proof the concept in a controlled clinical trial in healthy subjects, whether methylnaltrexone antagonizes the loperamide induced delay of oro-cecal and whole-gut transit time after oral administration of immediate and extended release capsules in comparison to subcutaneous administration.

Loperamide is an opioid agonist and acts on the µ-receptors in the myenteric plexus. It does not affect the central nervous system like other opioids. Loperamide significantly prolongs the mouth-to-cecum transit time as evaluated by the lactulose hydrogen breath test. This effect may be antagonized by the concomitant administration of naloxone.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 45 years
* sex: male and female
* ethnic origin: Caucasian
* minimal body weight: 62 kg
* body mass index: ≥ 19 kg/m² and ≤ 27 kg/m²
* good health as evidenced by the results of the clinical examination, ECG, and the laboratory check-up, which were judged by the clinical investigator not to differ in a clinical relevant way from the normal state
* written informed consent

Exclusion Criteria:

* hepatic and renal diseases and/or pathological findings, which might interfere with pharmacokinetics and pharmacodynamics of the study medication
* gastrointestinal diseases and/or pathological findings, which might interfere with pharmacokinetics and pharmacodynamics of the study medication
* drug or alcohol dependence
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day
* positive results in HIV, HBV and HCV screenings
* volunteers who were on a diet which could affect the pharmacokinetics of the drug
* heavy tea or coffee drinkers (more than 1 L per day)
* lactation, pregnancy test positive or not performed or women of child-bearing age without safe contraception
* volunteers suspected or known not to follow instructions of the clinical investigators
* volunteers who were unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they would have been exposed to as a result of their participation in the study
* volunteers liable to orthostatic dysregulation, fainting or blackouts
* participation in a clinical trial during the last 3 months prior to the start of the study
* less than 14 days after last acute disease
* less than 3 months after last blood donation
* any medication within 4 weeks prior to the intended first administration of the study medication which might have influenced functions of the gastrointestinal tract (e.g. laxatives, metoclopramide, loperamide, antacids, H2-receptor antagonists, proton pump inhibitors)
* any other medication within two weeks prior to the first administration of the study medication, but at least 10-time the half-live of the respective drug (except oral contraceptives)
* intake of grapefruit containing food or beverages within 14 days prior to administration of the study medication
* known allergic reactions to the active ingredients used or to constituents of the study medication
* deficiency of glucose-6-phosphate dehydrogenase

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Oro-cecal transit time | up to 24 h after administration of sulfasalazine
  Oro-cecal transit time (OCT) was defined as the first appearance of sulfapyridine in the blood after oral administration of 500 mg sulfasalazine immediate release tablets. Because of the high sensitivity of the analytical assay, the OCT was defined as the average of the times needed after sulfasalazine administration to exceed serum concentrations (cut-off) of 50 ng/ml (t50) and of 100 ng/ml (t100).
Average whole-gut transit time | up to 6 days after administration of methylnaltrexone
  Whole-gut transit time (WGT) was assessed by counting the appearance of radio-opaque markers of different shapes (Colon transit capsules) to different time pints in the stool, which were administered 24 h, 12 h and 1 h before administration of the methylnaltrexone study medication. The radio-opaque markers in the stool inside the sampling containers were visualized with an X-ray device (Philips Optimus, Philips Healthcare, Hamburg, Germany, CE 257303004) The images were stored and evaluated using the Agfa PACS Workstation, Impact-Version 5.2 (Agfa-Healthcare, Cologne, Germany).
renal clearances (CLR) | blood sampling at 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 12, 16, 24 h and urine sampling in 24 hours interval for 3 days after administration of methylnaltrexone
area under the concentrations-time curve (AUC) | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 12, 16, 24 h after administration of methylnaltrexone
maximum concentration (Cmax) | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 12, 16, 24 h after administration of methylnaltrexone
time of maximum concentration (Tmax) | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 12, 16, 24 h after administration of methylnaltrexone
terminal half-life (t1/2) | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 12, 16, 24 h after administration of methylnaltrexone
mean residence time (MRT) | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 12, 16, 24 h after administration of methylnaltrexone
distribution volume at steady-state (Vss) | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 12, 16, 24 h after administration of methylnaltrexone
total body clearance (CLtot) | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 12, 16, 24 h after administration of methylnaltrexone
relative bioavailability (F) | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 9, 10, 12, 16, 24 h after administration of methylnaltrexone
  Ratio AUC of IR and ER formulation over subcutaneous administration

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Ernst-Moritz-Arndt-University Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany